CLINICAL TRIAL: NCT03942315
Title: Recurrence of Hereditary Hemorrhagic Telangiectasia (HHT) After Liver Transplantation: Clinical Implications and Physiopathological Insights.
Brief Title: Recurrence of Hereditary Hemorrhagic Telangiectasia (HHT) After Liver Transplantation
Acronym: HHT
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: HHT
Record Dates: First submitted 2019-05-02; First posted 2019-05-08 (Actual); Last update posted 2019-05-08 (Actual); Status verified 2019-05

CONDITIONS: Hereditary Haemorrhagic Telangiectasia; Liver Transplant
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Liver transplant in Hereditary Hemorrhagic Telangiectasia: Hereditary Hemorrhagic Telangiectasia (HHT) patients who underwent a liver transplant in Lyon between 1993 and 2010, and who survived more than 1 year after transplantation.
  Interventions: Other: Data collection from standard follow-up after liver transplant

INTERVENTIONS:
Other: Data collection from standard follow-up after liver transplant — All patients underwent regular follow-up every 6 to 12 months after the first year post-liver transplant (LT). Complete laboratory investigations were performed at each visit. Doppler ultrasonography was performed every 1 to 3 years after LT. Computed tomography (CT) scan and/ or magnetic resonance imaging (MRI) was performed at 1, 5, 10, 15, and 20 years after LT, or when clinically indicated. All available radiological material was reviewed. Cardiac evaluation was performed regularly in patients who received transplant for cardiac failure.

SUMMARY:
Liver transplantation (LT) has been proposed as a curative treatment in hereditary hemorrhagic telangiectasia (HHT) with severe hepatic involvement. The investigating team provides a long-term evaluation of graft status after LT for HHT with a focus on the risk of recurrence. The present study included all patients prospectively followed up after LT for HHT in the Lyon Liver Transplant Unit from 1993 to 2010 with a survival of more than 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Hereditary Hemorrhagic Telangiectasia (HHT) patient who underwent liver transplant for HHT

Exclusion Criteria:

* Patient who died in the year following transplantation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hereditary Hemorrhagic Telangiectasia (HHT) patient who underwent liver transplant
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Change in graft status after liver transplant for Hereditary Haemorrhagic Telangiectasia (HHT) (risk of recurrence) | Every 6 months after transplantation up to 5 years
  Recurrent clinical examinations (including laboratory, histological and radiological investigations)

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme DUMORTIER, MD, Principal Investigator — Hospices Civils de Lyon (Hôpital Edouard Herriot )